CLINICAL TRIAL: NCT06720285
Title: The Efficacy of Regional Scalp Block Local Anesthesia as Preemptive Analgesia in Craniotomy Surgery
Brief Title: The Efficacy of Regional Scalp Block in Craniotomy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Dr. Soetomo Hospital, Surabaya (Unknown); Kementerian Riset dan Teknologi / Badan Riset dan Inovasi Nasional, Indonesia (Other Government)
Responsible Party: Principal Investigator, Dr. Christijogo Soemartono Waloejo, MD, Ph.D, Universitas Airlangga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB: 0769/KEPK/IX/2023; INA-XOYLZRE (Registry Identifier: The Indonesia Clinical Research Registry)
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Scalp Nerve Block; Craniotomy Surgery
Keywords: Regional anesthesia; Scalp Nerve Block; Craniotomy; Surgery
MeSH Terms: interventions — Nerve Block; Ropivacaine; Anesthesia, General; Analgesics, Opioid; Fentanyl; Propofol; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Treatment with Scalp Nerve Block (Experimental): General anesthesia induction was performed by administering fentanyl 1-2 mcg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg. Subsequently, scalp nerve block was performed with 0.5% ropivacaine.
  During surgery, a sudden rise of heart rate and blood pressure higher than 20% from baseline was considered as pain, and a bolus of fentanyl was administered as rescue analgesia.
  Interventions: Procedure: nerve block with 0.5% ropivacaine; Drug: General anesthesia and opioids (fentanyl, propofol, rocuronium)
- Standard Treatment (Active Comparator): General anesthesia induction was performed by administering fentanyl 1-2 mcg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg. Then, continuous fentanyl infusion as analgesia maintenance as the standard treatment. During surgery, a sudden rise of heart rate and blood pressure higher than 20% from baseline was considered as pain, and a bolus of fentanyl was administered as rescue analgesia.
  Interventions: Drug: General anesthesia and opioids (fentanyl, propofol, rocuronium)

INTERVENTIONS:
Procedure: nerve block with 0.5% ropivacaine — Compared to active comparator arm, the experimental arm received the same procedure except in the analgesia maintenance which was performed by nerve block of the scalp using 0.5% ropivacaine. However, during craniotomy surgery, pain may occur in patients in any arms. This was defined as a sudden rise of heart rate and blood pressure higher than 20% from baseline. In that case, a bolus of fentanyl was administered as rescue analgesia.
  Arms: Standard Treatment with Scalp Nerve Block
Drug: General anesthesia and opioids (fentanyl, propofol, rocuronium) — Compared to experimental arm, the active comparator arm received the same procedure except in the analgesia maintenance which was performed through continuous fentanyl infusion. However, during craniotomy surgery, pain may occur in patients in any arms. This was defined as a sudden rise of heart rate and blood pressure higher than 20% from baseline. In that case, a bolus of fentanyl was administered as rescue analgesia.

SUMMARY:
The objective of this clinical trial is to evaluate the role of scalp nerve block in craniotomy. The primary questions it seeks to answer are: What are the efficacy and safety profiles of scalp nerve block in craniotomy? The anesthesia protocol and monitoring were standardized for all participants. Participants were divided into two groups: the scalp nerve block group and the general anesthesia group. General anesthesia was induced using fentanyl (1-2 mcg/kg), propofol (1-2 mg/kg), and rocuronium (0.6 mg/kg). In the scalp nerve block group, a nerve block was administered using 0.5% ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years
* American Society of Anesthesiologists (ASA) classification I-III
* Glasgow Coma Scale (GCS) score ≥ 13
* Elective craniotomy

Exclusion Criteria:

- Patients with cardiovascular abnormalities, impaired renal and hepatic function, diabetes mellitus, systemic and/or scalp local infection, and those with a history of current dexamethasone administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | From enrollment until 24 hours post craniotomy surgery.
  Opioid used was fentanyl, and it was administered during and post surgery which was measured μg/kg.

SECONDARY OUTCOMES:
Pain Scale | 0 to 24 hours after surgery
  Pain scale was assessed using the Critical-care Pain Observational Tool (CPOT) every 4 hours
Laboratory Markers | After induction of anesthesia, 6 hours after incision, and 24 hours after surgery.
  Laboratory markers measured were Interleukin (IL)-6 (pg/mL), Tumor Necrosis Factor (TNF)-α (pg/mL), prostaglandin E2 (PGE2) (pg/mL), cortisol level (μg/dL), blood glucose level (mg/dL), neutrophil count (cells/μL), lymphocyte count (cells/μL) and neutrophil-to-lymphocyte ratio (NLR).
The patients with PONV | 0 to 24 hour after surgery
  Postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Christijogo Soemartono Waloejo, MD, Ph.D, Principal Investigator — Anesthesiology and Reanimation Department, Dr. Soetomo General Hospital, Universitas Airlangga, Indonesia
Locations (1):
- Dr. Soetomo Hospital, Surabaya, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The individual data may be requested through formal and reasonable request. This must be adressed to the principal investigator, and the decision is at his discretion.

REFERENCES:
- [Background] Chen Y, Ni J, Li X, Zhou J, Chen G. Scalp block for postoperative pain after craniotomy: A meta-analysis of randomized control trials. Front Surg. 2022 Sep 26;9:1018511. doi: 10.3389/fsurg.2022.1018511. eCollection 2022. PMID 36225222
- [Background] Costello TG, Cormack JR. Anaesthesia for awake craniotomy: a modern approach. J Clin Neurosci. 2004 Jan;11(1):16-9. doi: 10.1016/j.jocn.2003.09.003. No abstract available. PMID 14642359
- [Background] Benyahia NM, Verster A, Saldien V, Breebaart M, Sermeus L, Vercauteren M. Regional anaesthesia and postoperative analgesia techniques for spine surgery - a review. Rom J Anaesth Intensive Care. 2015 Apr;22(1):25-33. PMID 28913452
- [Background] Vadivelu N, Kai AM, Tran D, Kodumudi G, Legler A, Ayrian E. Options for perioperative pain management in neurosurgery. J Pain Res. 2016 Feb 10;9:37-47. doi: 10.2147/JPR.S85782. eCollection 2016. PMID 26929661
- [Background] Ghai B, Jafra A, Bhatia N, Chanana N, Bansal D, Mehta V. Opioid sparing strategies for perioperative pain management other than regional anaesthesia: A narrative review. J Anaesthesiol Clin Pharmacol. 2022 Jan-Mar;38(1):3-10. doi: 10.4103/joacp.JOACP_362_19. Epub 2022 Feb 4. PMID 35706649
- [Background] Gottschalk A, Berkow LC, Stevens RD, Mirski M, Thompson RE, White ED, Weingart JD, Long DM, Yaster M. Prospective evaluation of pain and analgesic use following major elective intracranial surgery. J Neurosurg. 2007 Feb;106(2):210-6. doi: 10.3171/jns.2007.106.2.210. PMID 17410701